CLINICAL TRIAL: NCT05932121
Title: The Effect of Postoperative Quality of Life and Cosmetic Result Between PTC Patients Underwent Thyroid Lobectomy Via Different Surgical Approach, Trans-axillary Approach vs Open Approach: A Cross-sectional Research
Brief Title: Cross-sectional Case and Control Study on Quality of Life, Appearance and Functions in PTC Via Different Surgical Approach
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: K4107-K23C1755
Record Dates: First submitted 2023-06-24; First posted 2023-07-06 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-06

CONDITIONS: Papillary Thyroid Carcinoma; Thyroid Cancer
Keywords: Papillary thyroid carcinoma; Surgical approaches; Voice assessment; Swallowing assessment; Cosmetic outcomes; Quality of life
MeSH Terms: conditions — Thyroid Cancer, Papillary; Thyroid Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PTC patients underwent thyroid lobectomy via trans-axillary approach: Case: PTC patients underwent thyroid lobectomy via trans-axillary approach.
  Interventions: Procedure: Thyroid lobectomy via trans-axillary approach
- PTC patients underwent thyroid lobectomy via open approach: Controls: PTC patients underwent thyroid lobectomy via open approach.
  Interventions: Procedure: Thyroid lobectomy via open approach

INTERVENTIONS:
Procedure: Thyroid lobectomy via trans-axillary approach — Patient with PTC underwent thyroid lobectomy via trans-axillary approach
  Groups: PTC patients underwent thyroid lobectomy via trans-axillary approach
Procedure: Thyroid lobectomy via open approach — Patient with PTC underwent thyroid lobectomy via open approach
  Groups: PTC patients underwent thyroid lobectomy via open approach

SUMMARY:
An observational cross-sectional case-control study on the postoperative quality of life (5 aspects, general quality of life, thyroid specific quality of life, scar appearance, voice and swallowing functions) of papillary thyroid carcinoma (PTC) patients underwent thyroid lobectomy via different approach, open vs trans-axillary. The patients are recruited in Peking Union Medical College Hospital (PUMCH) from 2020 to 2023 and are evaluated by follow-up with both outpatient visits and questionnaires made up of 9 validated scales.

DETAILED DESCRIPTION:
Thyroid carcinoma is the most common thyroid tumor with a rising incidence. By 2015, it has risen to the fourth most common tumor among all tumors in female. Papillary thyroid carcinoma (PTC), representing up to 80% of all thyroid carcinomas, mostly occurring in female between 30-50 years old, although it has an excellent long-term survival outcome, still it brings the patients concerns and complaints of the obvious scars left on their necks by operations via traditional open approach. Cosmetic approaches of thyroid surgery have been developing rapidly in the last two decades, through approaches including trans-axillary, transoral, and trans-breast-chest, thyroid operations are able to avoid leaving surgical scars on the necks and instead leaving them on other parts of bodies covering by clothes. However, concerns of this new emerging technique including its excision extent, surgical complication, clinical outcome, functional outcome and postoperative quality of life still remain unsolved. Well-matched, high quality-studies focused on functional outcomes, cosmetic outcomes, and quality of life with large samples are still missing.

This observational cross-sectional case-control study with follow-up on the postoperative quality of life, clinical outcomes, functional outcomes and cosmetic outcomes of PTC patients underwent thyroid lobectomy via different approach, open vs trans-axillary, aims on achieving comprehensive understanding on how different surgical approaches affect the quality of life, clinical outcomes and functional outcomes. Patients are recruited in PUMCH from 2020-2023 who underwent thyroid lobectomy and with a definite pathological diagnosis of PTC. Cases are defined as PTC patients who underwent thyroid lobectomy via trans-axillary approach. Controls are defined as PTC patients who underwent thyroid lobectomy via open approach. Controls are matched to cases with a 1:1 ratio according to gender, age, main operator.

The postoperative quality of life, functional outcomes will be evaluated by a questionnaire made up of 4 validated scales (EORTC thyroid cancer specific quality of life questionnaire (THY34-QoL); patient scar assessment questionnaire (PSAQ); voice handicap index questionnaire (VHI-10); Swallowing impairment score (SIS-6). Clinical outcomes will be evaluated by data collected both from inpatient medical records and outpatient follow-up medical records. To our knowledge, this is the largest PTC thyroid lobectomy via trans-axillary approach case-control study worldwide, the first study with the design of assigning control matched to cases by applying pre-matching score method in this field, and the first study to concentrate on both clinical outcomes and comprehensive postoperative quality of life including physical, functional, and cosmetic outcomes in PTC patients via different surgical approaches.

ELIGIBILITY:
Inclusion Criteria:

* PTC patients underwent thyroid lobectomy with pathological diagnosis of PTC after surgery

Exclusion Criteria:

* Refusal to participate; Patients with invalid or incomplete questionnaire results; Patients with another primary malignancy; Patients with severe immune disease or chronic disease accompanying with major organ failure.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All of the hospitalized patients of PTC with a definite pathological diagnosis who underwent thyroid lobectomy via trans-axillary approach and those who underwent thyroid lobectomy via open approach matched by age, gender and major operator with a ratio of 1: 1 from 2020 to 2023 in Peking Union Medical College Hospital.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-06-25 (Estimated); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Cosmetic outcomes | up to 3 years after surgery
  The primary outcome will be evaluated by scores of cosmetic outcomes of PTC patients underwent thyroid lobectomy via different surgical approach up to 3 years after surgery. The scores are evaluated by a follow-up questionnaire made up of cosmetic outcome via scale of PSAQ. Scores will be compared in case and control groups. Lower scores in PSAQ indicate poorer outcomes in this field.

SECONDARY OUTCOMES:
Thyroid cancer specific postoperative quality of life | up to 3 years after surgery
  The thyroid cancer specific postoperative quality of life will be evaluated by scores of thyroid cancer specific quality of life of PTC patients underwent thyroid lobectomy via different surgical approach up to 3 years after surgery. The scores are evaluated by a follow-up questionnaire made up of EORTC THY34-QoL scale. Scores will be compared in case and control groups. Higher scores in EORTC THY34-QoL indicate better quality of life.
Voice outcomes | up to 3 years after surgery
  The voice outcomes will be evaluated by scores of voice outcomes of PTC patients underwent thyroid lobectomy via different surgical approach up to 3 years after surgery. The scores are evaluated by a follow-up questionnaire made up of VHI-10 scale. Scores will be compared in case and control groups. Lower scores in VHI-6 indicate poorer outcomes in this field.
Swallowing function outcomes | up to 3 years after surgery
  The swallowing function outcomes will be evaluated by scores of swallowing function outcome of PTC patients underwent thyroid lobectomy via different surgical approach up to 3 years after surgery. The scores are evaluated by a follow-up questionnaire made up of SIS-6 scale. Scores will be compared in case and control groups. Lower scores in SIS-6 indicate poorer outcomes in swallowing function.
Time to recurrence | up to 3 years after surgery
  The time from the surgery to the recurrence (from date of surgery until the date of first documented recurrence including local recurrence, lymph node recurrence and distant metastasis).

CONTACTS AND LOCATIONS:
Overall Officials: Quan Liao, M.D, Study Chair — Department of General Surgery, Peking Union Medical College Hospital
Locations (1):
- Department of General Surgery, Peking Union Medical College Hospital, Peking Union Medical College & Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No